CLINICAL TRIAL: NCT06175013
Title: Prospective, Monocentric, Randomized, "Evaluator Blinded" Clinical Investigation to Evaluate the Efficacy and Safety of a Combination of Two Medical Devices and One Device Use in the Treatment of Toenail Onychomycosis
Brief Title: Evaluation of a Combination of Two Medical Devices and One Device Use in the Treatment of Toenail Onychomycosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Footcare Laboratories - Poderm Professional (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23E2000
Record Dates: First submitted 2023-11-28; First posted 2023-12-18 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Onychomycosis
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 : Sérum Mycose des ongles PURIFIANT (Experimental): Participant will apply Sérum PURIFIANT on the affected toenail, twice daily during the 112 days of the study.
  Interventions: Device: Sérum PURIFIANT
- Group 2 : Sérum Mycose des onglesPURIANT associated with Sérum Mycose des ongles BOOSTER (Experimental): Participant will apply Sérum PURIFIANT on the affected toenail, twice daily during the 112 days of the study.
  They will also apply Sérum BOOSTER, twice weekly before the Sérum PURIFIANT.
  Interventions: Device: Sérum PURIFIANT in association Sérum BOOSTER

INTERVENTIONS:
Device: Sérum PURIFIANT — Application of Sérum PURIFIANT only, twice daily during 112 days
  Arms: Group 1 : Sérum Mycose des ongles PURIFIANT
Device: Sérum PURIFIANT in association Sérum BOOSTER — Application of Sérum PURIFIANT twice daily during 112 days AND Application of Sérum BOOSTER before the Serum PURIFIANT, twice weekly
  Arms: Group 2 : Sérum Mycose des onglesPURIANT associated with Sérum Mycose des ongles BOOSTER

SUMMARY:
The goal of this clinical investigation is to evaluate the efficacy of the tested products in medium to moderate onychomycosis after 112 days of treatments.

The main question it aims to answer is the effectiveness of the use of a combination of two investigational devices (Sérum PURIFIANT + Sérum BOOSTER) on the percentage of healthy nail surface after 112 days of treatment.

Participants will apply one or two devices on the affected toenail during the study.

* Patients included on the groupe 1 will use Sérum PURIFIANT only, twice daily.
* Patient included on group 2 will use Sérum PURIFIANT, twice daily associated with Sérum BOOSTER twice weekly.

For this investigation, 44 patients (22 patients per group) presenting at least one infected toenail will be included to reach this objective.

DETAILED DESCRIPTION:
Onychomycosis is a fungal infection of the nail apparatus that causes discoloration, thickening, and separation from the nail bed.

It is primarily caused by dermatophytes, which are infectious fungi that feed on the keratin present in the skin, hair and nails. Onychomycosis has several clinical presentations, including distal and lateral subungual onychomycosis which is the most common form, proximal subungual onychomycosis, superficial white onychomycosis, and total dystrophic onychomycosis.

Onychomycosis affects toenails more often than fingernails because of their slower growth, reduced blood supply, and frequent confinement in dark, moist environments. (1) The severity of onychomycosis can be described as mild, moderate, or severe. Published studies will assign a label of mild-moderate disease if less than approximately 60% of the nail is showing symptoms.

Onychomycosis is the most common nail infection worldwide occurring in 10% of the general population but is more common in older adults. Despite treatment, the recurrence rate of onychomycosis is 10% to 50% as a result of reinfection or lack of mycotic cure.

Topical drugs for onychomycosis generally come in the form of lacquers or solutions directly applied to the surface of the nail.

The principal aim of this study is to evaluate the efficacy of the tested products in medium to moderate onychomycosis after 112 days of treatments. For this study, 44 patients (22 patients per group) presenting at least one infected toenail will be included to reach this objective.

ELIGIBILITY:
Inclusion Criteria:

* Patient having given freely her/his informed, written consent.
* Patient having a good general health.
* Age: more than 18 years.
* Patient cooperative and aware of the devices' modalities of use and the necessity and duration of the controls so that perfect adhesion to the protocol can be expected.
* Patient being psychologically able to understand information and to give his/her consent.
* Patient with nails superficial onychomycosis on at least one great toenail or light to moderate disto-lateral onychomycosis (without matrix involvement and involvement <2/3 of the tablet)
* Patient with slight to moderate impact of thickness of the nail and no deformation of the nail.
* Patient with slight to moderate impact of thickness of the nail and no deformation of the nail.
* Patient with positive KOH staining.
* Women of childbearing potential should use an accepted contraceptive regimen (to investigator's discretion) since at least 12 weeks before the beginning of the study, during all the study.

Exclusion Criteria:

* Pregnant or nursing woman or planning a pregnancy during the investigation.
* Patient considered by the investigator likely to be non-compliant with the protocol.
* Patient enrolled in another clinical trial during the test period.
* Patient having a known allergy or hypersensitivity to one of the constituents of the tested products.
* Patient with unstructured nail, severe microcracking or severe onycholysis.
* Patient with nails and nails contour with severe lesions
* Patient having used any systemic antifungal treatment in the last 6 months before inclusion.
* Patient having used any topical antifungal treatment in the last 3 months before inclusion.
* Patient with a condition or receiving a medication which, in the investigator's judgment, put the patient at undue risk.
* Patient suffering from serious or progressive diseases (to investigator's discretion) such as uncontrolled diabetes, peripheral circulatory disease, HIV, lichen planus, immunosuppressive pathology, chronic venous insufficiency, Peripheral Arterial Obstructive Disease, delay or lack of ungual growth …
* Patient with cutaneous pathology on studied zone (onychogryphosis, congenital ungual deformation, toe deformation or of the foot, Hallux Valgus, Hallux rigidus, Hallux extensus, toe claws or other pathologies than onychomycosis like angioma, dermatitis…).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of healthy surface | Day 0, Day 112
  The effect of the products on percentage of healthy surface will be evaluated at D112 by the mean variation from baseline in the group using a combination of two devices (Sérum PURIFIANT + Sérum BOOSTER).
  Evaluation is done in blind by digital analysis of photographs of the infected toenail.

SECONDARY OUTCOMES:
Percentage of healthy surface in group 1 | Day 0, Day 112
  The effect of the product on percentage of healthy surface will be evaluated at D112 by the mean variation from baseline in the group using only one device (Sérum PURIFIANT).
Percentage of healthy surface comparison | Day 0, Day 112
  The effect of the products on percentage of healthy surface will be evaluated at D112 by comparing mean variation from baseline between the two groups.
Onychomycosis | Day 0, Day 112
  The effect of the product on onychomycosis improvement will be evaluated at D0 and 112 days after treatment, on a scale from 0 normal to 3 severe.
  The effect of the products on clinical parameters will be evaluated by comparing mean variation from D0 within group and between the two groups.
Onycholysis | Day 0, Day 112
  The effect of the product on onycholysis improvement will be evaluated at D0 and 112 days after treatment, on a scale from 0 normal to 3 severe The effect of the products on clinical parameters will be evaluated by comparing mean variation from D0 within group and between the two groups.
Nail microcacking | Day 0, Day 112
  The effect of the product on nail microcacking improvement will be evaluated at D0 and 112 days after treatment. Number of nail microcracking will be collected.
  The effect of the products on clinical parameters will be evaluated by comparing mean variation from D0 within group and between the two groups.
Nail opacity | Day 0, Day 112
  The effect of the product on nail opacity improvement will be evaluated at D0 and 112 days after treatment, on a scale from 0 transparent to 4 Very opaque The effect of the products on clinical parameters will be evaluated by comparing mean variation from D0 within group and between the two groups.
KOH staining | Day 0, Day 112
  Percentage of patients with positive KOH staining at the screening visit and 112 days after treatment in each group and compared between the two groups.
QoL | Day 0, Day 112
  Percentage of patient with an improvement of their quality of life (QoL) by analysis of NailQoL patient answers at D0 and 112 days after treatment in each group and compared between the two groups.
Patient questionnaire | Day 0, Day 112
  Analysis of the answers to the patient questionnaire regarding effectiveness, tolerance, and acceptability of the investigational devices 112 days after treatment in each group. Answer will be on a scale from Totally agree to totally disagree
Tolerance | Day 0, Day 112
  Products tolerance will be assessed by the investigator and the patient at D112 on a 4 points scale from verry bad tolerance to very good tolerance
Adverse event | Screening visit, Day 0, Day 112
  Products safety will be assessed by collection of Adverse Events (AEs) throughout the study. AEs will be summarized and tabulated by severity, causality, action taken and outcome, using descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Aslham DOARIKA, Principal Investigator — Insight Research

IPD SHARING:
Plan to Share IPD: No